CLINICAL TRIAL: NCT06347003
Title: Double-blind, Placebo-controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Plozasiran in Adults With Severe Hypertriglyceridemia
Brief Title: Study of Plozasiran (ARO-APOC3) in Adults With Severe Hypertriglyceridemia
Acronym: SHASTA-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROAPOC3-3003; 2023-509300-14 (EudraCT Number)
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Severe Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — plozasiran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Plozasiran Injection (Experimental): 4 doses of plozasiran (ARO-APOC3) by subcutaneous (sc) injection
  Interventions: Drug: Plozasiran Injection
- Placebo (Placebo Comparator): calculated volume to match active treatment by sc injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Plozasiran Injection — ARO-APOC3 Injection
  Other Names: ARO-APOC3
  Arms: Plozasiran Injection
Drug: Placebo — sterile normal saline (0.9% NaCl)
  Arms: Placebo

SUMMARY:
This Phase 3 study will evaluate the safety and efficacy of plozasiran injection (ARO-APOC3) in adult participants with severe hypertriglyceridemia (SHTG). After providing informed consent eligible participants will be randomized to receive 4 doses (once every 3 months) of plozasiran or placebo, and be evaluated for efficacy and safety. After month 12, eligible participants will be offered an opportunity to continue in an optional open-label extension under a separate protocol.

ELIGIBILITY:
Inclusion Criteria:

* Males, or nonpregnant (who do not plan to become pregnant) nonlactating females, who are ≥18 years of age at screening
* Established diagnosis of severe hypertriglyceridemia (SHTG) and prior documented evidence (medical history) of fasting TG levels of ≥ 500 mg/dL (≥5.65mmol/L)
* Mean fasting TG level ≥500 mg/dL (≥5.65 mmol/L) collected at 2 separate and consecutive visits at least 7 days apart and no more than 17 days apart during the screening period
* Fasting low density lipoprotein-cholesterol (LDL-C) ≤130 mg/dL (≤3.37 mmol/L) at screening
* Screening HbA1C ≤9.0%
* Willing to follow diet counseling and maintain a stable low-fat diet
* Must be on standard of care lipid and TG lowering medications per local guidelines (unless documented as intolerant as determined by the Investigator, including an inability to safely administer or re-administer a specific drug because of fear, preference, genetic, clinical, or metabolic considerations, or due to a previous adverse reaction associated with, attributed to, or caused by specific drug)

Exclusion Criteria:

* Use of any hepatocyte-targeted small interfering ribonucleic acid (siRNA) that targets lipids and/or triglycerides within 365 days before Day 1 (except inclisiran, which is permitted). Administration of investigational drug and inclisiran must be separated by at least 4 weeks
* Use of any other hepatocyte-targeted siRNA or antisense oligonucleotide molecule within 60 days or within 5-half-lives before Day 1 based on plasma pharmacokinetics (PK), whichever is longer
* Known diagnosis of familial chylomicronemia syndrome (FCS) (type 1 Hyperlipoproteinemia) by documentation of confirmed homozygote or double heterozygote for loss-of-function mutations in type 1-causing genes
* Acute pancreatitis within 4 weeks prior to screening
* Body mass index >45kg/m^2

Note: Additional Inclusion/Exclusion criteria may apply per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Fasting Serum Triglyceride (TG) Levels from Baseline to Month 12 Compared to Placebo | Baseline, Month 12

SECONDARY OUTCOMES:
Percent Change in Fasting Serum TG Levels from Baseline to Month 10 Compared to Placebo | Baseline, Month 10
Proportion of Participants Who Achieve Fasting TG Levels of <500 mg/dL (<5.65 mmol/L) at Month 12 Compared to Placebo | Baseline, Month 12
Proportion of Participants Who Achieve Fasting TG Levels of <150 mg/dL (<1.69 mmol/L) at Month 12 Compared to Placebo | Baseline, Month 12
Percent change in remnant cholesterol (VLDL-C) from baseline to Month 12 compared to placebo | Baseline, Month 12
Percent change in non-HDL-C from baseline to Month 12 compared to placebo | Baseline, Month 12
Adjudicated AP Event Rate During the Treatment Period Compared to Placebo From Day 1 to Month 12 | Month 12
Number of participants with adverse events (AEs) and serious adverse events (SAEs) over time through Month 12 as compared to placebo | From first dose of study drug through Month 12
Incidence Rates of New-Onset Diabetes Mellitus (NODM) Throughout the Course of Treatment | From first dose of study drug through Month 12
Incidence rates of impaired glucose tolerance throughout the course of treatment | From first dose of study drug through Month 12
Incidence rates of worsening of existing diabetes throughout the course of treatment | From first dose of study drug through Month 12
Change from baseline in HbA1c during the treatment period compared to placebo. | From first dose of study drug through Month 12
Change from Baseline in Fasting Blood Glucose During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Change from Baseline in C-peptide During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Change from Baseline in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Change from Baseline in Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related Adverse Events (TRAEs) Associated with Worsening Glycemic Control During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Initiation of New Medication for Hyperglycemia Among Study Participants Not Known to Have Pre-existing Diabetes Mellitus During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Adjudicated Major Adverse Cardiovascular Events (MACE) Rates During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Incidence of Anti-drug Antibodies (ADA) to Plozasiran in Participants Receiving Plozasiran Over Time Through Month 12 | From first dose of study drug through Month 12
Titers of Anti-drug Antibodies (ADA) to Plozasiran in Participants Receiving Plozasiran Over Time Through Month 12 | From first dose of study drug through Month 12
Change and/or percent change from baseline to Month 12 in liver fat content using MRI-PDFF, only in a subset of subjects | Baseline, Month 12

CONTACTS AND LOCATIONS:
Locations (196):
- United States (52):
  - Research Center 1, Garden Grove, California
  - Research Center 2, Lake Forest, California
  - Research Center 3, Montclair, California
  - Research Center 4, Panorama City, California
  - Research Center 5, Redding, California
  - Research Center 6, Colorado Springs, Colorado
  - Research Center 7, Hialeah, Florida
  - Research Center 8, Lake City, Florida
  - Research Center 9, Miami Lakes, Florida
  - Research Center 10, Mt. Dora, Florida
  - Research Center 11, Orlando, Florida
  - Research Center 12, Pensacola, Florida
  - Research Center 13, Tamarac, Florida
  - Research Center 14, Tampa, Florida
  - Research Center 15, Macon, Georgia
  - Research Center 16, Savannah, Georgia
  - Research Center 17, Park Ridge, Illinois
  - Research Center 18, Eunice, Louisiana
  - Research Center 19, Baltimore, Maryland
  - Research Center 20, Flint, Michigan
  - Research Center 21, Minneapolis, Minnesota
  - Research Center 22, Olive Branch, Mississippi
  - Research Center 23, Jefferson City, Missouri
  - Research Center 24, St Louis, Missouri
  - Research Center 26, Omaha, Nebraska
  - Research Center 25, Omaha, Nebraska
  - Research Center 27, Las Vegas, Nevada
  - Research Center 29, Long Island City, New York
  - Research Center 30, New York, New York
  - Research Center 31, Rochester, New York
  - Research Center 28, The Bronx, New York
  - Research Center 32, Vestal, New York
  - Research Center 33, Morehead City, North Carolina
  - Research Center 34, Winston-Salem, North Carolina
  - Research Center 35, Cincinnati, Ohio
  - Research Center 36, Columbus, Ohio
  - Research Center 37, Norman, Oklahoma
  - Research Center 38, Oklahoma City, Oklahoma
  - Research Center 39, Powell, Tennessee
  - Research Center 40, El Paso, Texas
  - Research Center 47, Houston, Texas
  - Research Center 45, Houston, Texas
  - Research Center 46, Houston, Texas
  - Research Center 42, Houston, Texas
  - Research Center 44, Houston, Texas
  - Research Center 43, Houston, Texas
  - Research Center 41, Houston, Texas
  - Research Center 48, Laredo, Texas
  - Research Center 49, Missouri City, Texas
  - Research Center 50, Plano, Texas
  - Research Center 51, San Antonio, Texas
  - Research Center 52, Seattle, Washington
- Argentina (10):
  - Research Center 8, Ramos Mejía, Buenos Aires
  - Research Center 10, San Isidro, Buenos Aires
  - Research Center 7, Temperley, Buenos Aires
  - Research Center 4, Córdoba, Córdoba Province
  - Research Center 9, Córdoba, Córdoba Province
  - Research Center 5, Córdoba, Córdoba Province
  - Research Center 3, Córdoba, Córdoba Province
  - Research Center 6, Buenos Aires
  - Research Center 2, Buenos Aires
  - Research Center 1, Buenos Aires
- Australia (7):
  - Research Center 1, Blacktown, New South Wales
  - Research Center 4, Concord, New South Wales
  - Research Center 5, Merewether, New South Wales
  - Research Center 2, Box Hill, Victoria
  - Research Center 7, Clayton, Victoria
  - Research Center 3, Heidelberg, Victoria
  - Research Center 6, Crawley, Western Australia
- Belgium (6):
  - Research Center 4, Gozée
  - Research Center 6, Hasselt
  - Research Center 3, Mechelen
  - Research Center 2, Namur
  - Research Center 5, Roeselare
  - Research Center 1, Wetteren
- Brazil (14):
  - Research Center 10, Vitória, Espírito Santo
  - Research Center 12, Salvador, Estado de Bahia
  - Research Center 13, Salvador, Estado de Bahia
  - Research Center 14, Salvador, Estado de Bahia
  - Research Center 5, Belo Horizonte, Minas Gerais
  - Research Center 8, Campina Grande do Sul, Paraná
  - Research Center 2, Curitiba, Paraná
  - Research Center 4, Belém, Pará
  - Research Center 6, Porto Alegre, Rio Grande do Sul
  - Research Center 9, Porto Alegre, Rio Grande do Sul
  - Research Center 1, Campinas, São Paulo
  - Research Center 7, São Paulo, São Paulo
  - Research Center 11, São Paulo, São Paulo
  - Research Center 3, Votuporanga, São Paulo
- Bulgaria (15):
  - Research Center 8, Burgas, Burgas
  - Research Center 11, Rousse, Ruse
  - Research Center 15, Sofia, Sofia
  - Research Center 7, Sofia, Sofia
  - Research Center 12, Blagoevgrad
  - Research Center 10, Kardzhali
  - Research Center 1, Pleven
  - Research Center 3, Pleven
  - Research Center 4, Plovdiv
  - Research Center 2, Plovdiv
  - Research Center 9, Plovdiv
  - Research Center 13, Sofia
  - Research Center 6, Sofia
  - Research Center 5, Sofia
  - Research Center 14, Sofia
- Canada (8):
  - Research Center 3, Victoria, British Columbia
  - Research Center 1, Brampton, Ontario
  - Research Center 8, London, Ontario
  - Research Center 2, Sarnia, Ontario
  - Research Center 5, Waterloo, Ontario
  - Research Center 6, Montreal, Quebec
  - Research Center 4, Québec, Quebec
  - Research Center 7, Halifax
- China (23):
  - Research Center 11, Bengbu, Anhui
  - Research Center 23, Beijing, Beijing Municipality
  - Research Center 22, Beijing, Beijing Municipality
  - Research Center 7, Guangzhou, Guangdong
  - Research Center 19, Guanzhou, Guangdong
  - Research Center 8, Liuchow, Guangxi Zhuang
  - Research Center 13, Xingtai, Hebei
  - Research Center 6, Luoyang, Henan
  - Research Center 21, Wuhan, Hubei
  - Research Center 4, Changsha, Hunan
  - Research Center 18, Changsha, Hunan
  - Research Center 16, Baotou, Inner Mongolia
  - Research Center 10, Suzhou, Jiangsu
  - Research Center 9, Shanghai, Shanghai Municipality
  - Research Center 12, Shanghai, Shanghai Municipality
  - Research Center 2, Yuncheng, Shanxi
  - Research Center 17, Chengdu, Sichuan
  - Research Center 20, Tianjin, Tianjin Municipality
  - Research Center 1, Beijing, Xicheng
  - Research Center 15, Wenzhou, Zhejiang
  - Research Center 5, Hangzhou
  - Research Center 3, Liaocheng
  - Research Center 14, Nanchang
- Croatia (4):
  - Research Center 1, Zagreb, City of Zagreb
  - Research Center 2, Krapinske Toplice
  - Research Center 3, Zagreb
  - Research Center 4, Zagreb
- Czechia (9):
  - Research Center 8, Prague, Prague
  - Research Center 4, Prague, Prague
  - Research Center 3, Hodonín
  - Research Center 6, Hradec Králové
  - Research Center 1, Ostrava
  - Research Center 7, Praha 1-Nove Mesto
  - Research Center 5, Praha 4-Krc
  - Research Center 2, Uherské Hradiště
  - Research Center 9, Ústí nad Labem
- Hungary (6):
  - Research Center 1, Budapest
  - Research Center 4, Budapest
  - Research Center 2, Budapest
  - Research Center 6, Budapest
  - Research Center 3, Szeged
  - Research Center 5, Veszprém
- Italy (6):
  - Research Center 3, Rozzano, Milano
  - Research Center 2, Palermo, Sicily
  - Research Center 6, Bologna
  - Research Center 5, Brescia
  - Research Center 4, Milan
  - Research Center 1, Roma
- Poland (12):
  - Research Center 15, Żarów, Swidnica
  - Research Center 7, Bydgoszcz
  - Research Center 11, Elblag
  - Research Center 10, Katowice
  - Research Center 13, Krakow
  - Research Center 17, Krakow
  - Research Center 8, Krakow
  - Research Center 12, Lodz
  - Research Center 18, Warsaw
  - Research Center 9, Warsaw
  - Research Center 16, Wroclaw
  - Research Center 14, Wroclaw
- Romania (9):
  - Research Center 3, Brasov, Brașov County
  - Research Center 1, Bucharest, București
  - Research Center 2, Cluj-Napoca, Cluj
  - Research Center 6, Alba Iulia, Jud. Alba
  - Research Center 4, Ploieşti, Jud. Prahova
  - Research Center 5, Timișoara, Timiș County
  - Research Center 8, Deva
  - Research Center 7, Galati
  - Research Center 9, Târgu Mureş
- Slovakia (6):
  - Research Center 4, Banská Bystrica, Banská Bystrica Region
  - Research Center 1, Košice, Košice Region
  - Research Center 3, Moldava nad Bodvou, Košice Region
  - Research Center 6, Bardejov
  - Research Center 5, Bratislava
  - Research Center 2, Žilina, Žilina Region
- Spain (4):
  - Research Center 2, Barcelona
  - Research Center 3, Barcelona
  - Research Center 1, Valencia
  - Research Center 4, Zaragoza
- United Kingdom (5):
  - Research Center 3, Torpoint, Cornwall
  - Research Center 5, Torquay, Devon
  - Research Center 2, Plymouth, Devpn
  - Research Center 1, London
  - Research Center 4, London

IPD SHARING:
Plan to Share IPD: No